CLINICAL TRIAL: NCT04331249
Title: Perioperative Management Evaluation in Patients With Implanted Cardiac Electronic Devices
Brief Title: Perioperative Management Evaluation in Patients With CIED
Acronym: EVINCE
Status: Recruiting | Type: Observational
Sponsor: Klinikum-Fuerth (Other)
Collaborators: Klinikum Nürnberg (Other)
Responsible Party: Sponsor
Other Study IDs: EVINCE_KHF
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Pacemaker Malfunction; ICD Malfunction; Cardiac Pacemaker Electrical Interference; Anesthesia Complication; Surgery--Complications
Keywords: pacemaker; implanted cardioverter defibrillator; cardiac resynchronisation therapy; management, peri-operative
MeSH Terms: interventions — Surgical Procedures, Operative; Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery or catheter based cardiac procedure (catheter ablation) — patients with implanted CIED (pacemaker, ICD or CRT) that undergo any surgery or any catheter based cardiac procedure (e.g. radiofrequency ablation)

SUMMARY:
Background: Recommendations for peri-operative management in patients with implanted cardiac electronic devices (CIED) are often based on older data from case reports and small collectives.

Objective: To evaluate the peri-operative management and outcome of patients with implanted CIED undergoing non-CIED related surgery or catheter-interventional procedures in clinical routine.

Study design: bi-center, non-randomized, observational registry, retrospective data-collection, on-going prospective patient enrollment, descriptive statistics

Primary endpoint: number and type of peri-operative adverse device related events (ADE) Secondary endpoints: pre-interventional data (patient characteristics, data from CIED interrogation); peri-interventional data (type of surgery/intervention, anesthesiology techniques, any AE), postinterventional data (data from post-interventional CIED interrogation, need for reprogramming / device revision).

Inclusion criteria: implanted CIED, non-CIED related surgical or catheter-based intervention, peri-procedural CIED interrogation, age >18 years Exclusion criteria: no implanted CIED, no data from any peri-procedural CIED interrogation available

Patient enrollment: retrospectively beginning from 2008, further on-going prospective inclusion Sample size: For the observational study, there is no pre-specified sample size. Data from more than 500 patients undergoing > 700 interventions are expected.

DETAILED DESCRIPTION:
Background: The number of worldwide implanted cardiac electronic devices (CIED) is increasing continuously. On the other hand, the number of (more and more complex) surgical and catheter based interventions in this population is increasing as well. Recommendations for peri-operative management are often based on older data from case reports and small collectives. Data especially in particular subpopulations is limited.

Objective: The study aims to evaluate the peri-operative management and outcome of patients with implanted CIED undergoing non-CIED related surgery or catheter interventional procedures (ablation) in clinical routine. Data from the study are expected to provide evidence for recommendations improving perioperative management and device programming.

Study design: bi-center, non-randomized, observational registry, retrospective data-collection, on-going prospective patient enrollment, descriptive statistics Centers: Klinikum Fuerth (dep. for Heart and Lung disease, section for clinical electrophysiology), Klinikum Nuernberg (dep. for Heart surgery).

Patients and methods:

Primary endpoint: number and type of peri-operative adverse device related events (ADE)

- all complaints, adverse events and adverse device effects will be documented and classified according to the ISO/DIS 14155 - Clinical Investigation of medical Devices in Human Subjects - Good Clinical Practices with respect to their relationship to the surgical or catheter intervention and [Stark NJ. A New standard for medical device adverse event classification. J of Clinical Research Best Practices 2009; 5(12): 1-7].

Secondary endpoints: pre-interventional data (patient characteristics, data from CIED interrogation); peri-interventional data (type of surgery/intervention, anesthesiology techniques, any AE), post-interventional data (data from post-interventional CIED interrogation, need for reprogramming / device revision).

Subpopulations: cardiac surgery, vascular surgery, catheter ablation, ICD and mode of therapy inhibition, CRT, automatic features

Inclusion criteria:

patients with implanted CIED undergoing non-CIED related surgical or catheter-based procedure, peri-procedural CIED interrogation, age >18 years Exclusion criteria: no implanted CIED, no data from peri-procedural CIED interrogation available.

Patient enrollment: retrospectively from the clinical records beginning from 2008, further on-going prospective inclusion Data acquisition: Data will be collected in CRF´s from the patient's history, the computer based clinical information system / clinical records and data records from CIED interrogations

Sample size: For the observational study, there is no pre-specified sample size.

Data from more than 500 patients undergoing > 700 interventions are expected.

Data security: Study related data are collected by the study investigators in an anonymous clinic-internal data-base, that is password protected.

All investigators have to provide valid GCP training.

Risk estimation: the study is observational and descriptive with anonymized data collection/analysis and therefore adds no risk to the study population

ELIGIBILITY:
Inclusion Criteria:

* implanted CIED (e.g. pacemaker, ICD, CRT),
* performed (non-CIED related) surgical or catheter-based procedure,
* data from peri-procedural CIED interrogation available
* age >18 years

Exclusion Criteria:

* no implanted CIED,
* no data from any peri-interventional CIED interrogation available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment of all consecutive patients according to the inclusion criteria, undergoing surgery or catheter-ablation at the Klinikum Fuerth or Klinikum Nueremberg. Data collection will be
  * retrospectively beginning from 2008,
  * on-going with further prospective data collection and patient enrollment. If possible, patients will be enrolled at pre-interventional device interrogation. If there is no pre-interventional device interrogation (e.g. in case of urgent or emergency surgery), patients will be enrolled retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
surgery or catheter-based procedure related (S)ADE | 1 month post-procedural
  any (S)ADE related to the surgical or catheter-based procedure

SECONDARY OUTCOMES:
device: post-procedural pacing threshold increase | 1 month post-procedural
  post-procedural pacing threshold increase > 50% compared with the pre-procedural threshold (given a safety margin of 100%)
device: post-procedural sensing decrease | 1 month post-procedural
  post-procedural sensing decrease by > 50% compared with the pre-procedural sensing
device: post-procedural lead impedance | 1 month post-procedural
  post-procedural lead impedance is different by > 25% compared with the pre-procedural impedance

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bastian, MD, Principal Investigator — Klinikum Fuerth, European Society of Cardiology, European Heart Rhythm Society
Locations (2):
- Germany (2):
  - Klinikum Fuerth, Fürth, Bavaria
  - Klinikum Nuernberg, Nuremberg, Bavaria

IPD SHARING:
Plan to Share IPD: Undecided